CLINICAL TRIAL: NCT05767957
Title: The Contribution Of Cognitivo-Behavorial Therapy In Treatment Of Shoulder Apprehension: A Randomized Clinical Study
Brief Title: Contribution Of Cognitivo-Behavorial Therapy In Shoulder Apprehension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Epaule Coude CEPCO (Other)
Collaborators: Gregory Cunningham (Unknown); Alexandre Laedermann (Unknown); Benoît Borner (Unknown); Yannick Thilby (Unknown); Suzanne Gard (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-01912
Record Dates: First submitted 2022-07-25; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Shoulder Dislocation; Shoulder Instability
MeSH Terms: conditions — Shoulder Dislocation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Control group: rehabilitation physiotherapy by physiotherapist using conventional technique alone.
  Intervention group: rehabilitation physiotherapy by physiotherapist according to conventional technique, with the addition of techniques from cognitive-behavioral therapies.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: Rehabilitation physiotherapy
- Intervention group (Experimental)
  Interventions: Other: Cognitive-behavioral therapies in addition to rehabilitation physiotherapy

INTERVENTIONS:
Other: Rehabilitation physiotherapy — Rehabilitation physiotherapy by physiotherapist using conventional technique alone.
  Arms: Control group
Other: Cognitive-behavioral therapies in addition to rehabilitation physiotherapy — Rehabilitation physiotherapy by physiotherapist according to conventional technique, with the addition of techniques from cognitive-behavioral therapies.
  Arms: Intervention group

SUMMARY:
Randomized controlled double-blind study aimed at studying the contribution of cognitive-behavioral therapy in the treatment of shoulder apprehension. Comparison of 2 physiotherapy techniques in the context of shoulder instability.

Control group: rehabilitation physiotherapy by physiotherapist using conventional technique alone.

Intervention group: rehabilitation physiotherapy by physiotherapist according to conventional technique, with the addition of techniques from cognitive-behavioral therapies.

DETAILED DESCRIPTION:
Traumatic anterior instability of the shoulder is one of the most frequent lesions of the shoulder, the majority of cases of which occur in adolescents, with a risk of recurrence close to 90% if it occurs before the age of 20 years. It can be treated conservatively or surgically. Stabilizing surgery of the glenohumeral joint offers satisfactory results for people suffering from shoulder instability. Like subjects treated conservatively, patients undergoing stabilizing surgery remain apprehensive after the operation in 2 to 51% of cases. Currently, no rehabilitation program has demonstrated superior effectiveness, during instability treated conservatively or during postoperative rehabilitation. Recent studies have shown that cortical reorganization takes place, especially in areas of fear and anxiety. Faced with the need to develop physiotherapeutic management in post-traumatic unstable shoulder, this study aims to evaluate the contribution of cognitive-behavioral therapy, by including a neuropsychological axis in the rehabilitation of patients.

This study is randomized and controlled, multicenter, including 144 patients suffering from apprehension of the shoulder, divided into two treatment groups. Both groups will receive a conventional physiotherapy protocol including individual sessions and home exercises. The physiotherapists in the intervention group will also have received training in the use of techniques from Cognitive-Behavioral Therapies. Data will be collected before the introduction of physiotherapy, after 6, 12, 24 and 52 weeks of treatment. In the event of surgery, the data will also be collected preoperatively. The primary outcome is apprehension measured by the Rowe score. The secondary outcomes are apprehension measured by the apprehension and relocation tests, and the Tampa Scale for Kinesiophobia, as well as shoulder function, measured by the Simple Shoulder Test and the Subjective Shoulder Value.

ELIGIBILITY:
Inclusion Criteria:

* positive apprehension test;
* traumatic anterior dislocation of the glenohumeral joint requiring or not surgical stabilization according to Bankart or Latarjet;
* good oral and written comprehension of French;
* age between 15 and 45 years old.

Exclusion Criteria:

* associated tendon injury requiring surgical treatment;
* fracture other than Bankart fracture;
* multidirectional instability (MDI);
* peripheral neurological lesion in the upper limb;
* central neurological lesion;
* diagnosed psychosis, depression or epilepsy.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rowe score | enrolment
  Score for Shoulder Stability; 0-100 points (excellent: 90-100 pts; good: 75-89 pts; average: 51-74 pts; bad: <50 pts)
Rowe score | 6 weeks
  Score for Shoulder Stability; 0-100 points (excellent: 90-100 pts; good: 75-89 pts; average: 51-74 pts; bad: <50 pts)
Rowe score | 3 months
  Score for Shoulder Stability; 0-100 points (excellent: 90-100 pts; good: 75-89 pts; average: 51-74 pts; bad: <50 pts)
Rowe score | 6 months
  Score for Shoulder Stability; 0-100 points (excellent: 90-100 pts; good: 75-89 pts; average: 51-74 pts; bad: <50 pts)
Rowe score | 12 months
  Score for Shoulder Stability; 0-100 points (excellent: 90-100 pts; good: 75-89 pts; average: 51-74 pts; bad: <50 pts)

SECONDARY OUTCOMES:
Shoulder Range Of Motion: flexion | enrolment
  unit of measure: angle 0-180° degrees (worst: 0°; best: 180°); measurement tool: goniometer
Shoulder Range Of Motion: flexion | 3 months
  unit of measure: angle 0-180° degrees (worst: 0°; best: 180°); measurement tool: goniometer
Shoulder Range Of Motion: flexion | 6 months
  unit of measure: angle 0-180° degrees (worst: 0°; best: 180°); measurement tool: goniometer
Shoulder Range Of Motion: flexion | 12 months
  unit of measure: angle 0-180° degrees (worst: 0°; best: 180°); measurement tool: goniometer
Shoulder Range Of Motion: abduction | enrolment
  unit of measure: angle 0-180° degrees (worst: 0°; best: 180°); measurement tool: goniometer
Shoulder Range Of Motion: abduction | 3 months
  unit of measure: angle 0-180° degrees (worst: 0°; best: 180°); measurement tool: goniometer
Shoulder Range Of Motion: abduction | 6 months
  unit of measure: angle 0-180° degrees (worst: 0°; best: 180°); measurement tool: goniometer
Shoulder Range Of Motion: abduction | 12 months
  unit of measure: angle 0-180° degrees (worst: 0°; best: 180°); measurement tool: goniometer
Shoulder Range Of Motion: external rotation | enrolment
  unit of measure: angle 0-90° degrees (worst: 0°; best: 90°); measurement tool: goniometer
Shoulder Range Of Motion: external rotation | 3 months
  unit of measure: angle 0-90° degrees (worst: 0°; best: 90°); measurement tool: goniometer
Shoulder Range Of Motion: external rotation | 6 months
  unit of measure: angle 0-90° degrees (worst: 0°; best: 90°); measurement tool: goniometer
Shoulder Range Of Motion: external rotation | 12 months
  unit of measure: angle 0-90° degrees (worst: 0°; best: 90°); measurement tool: goniometer
Shoulder Range Of Motion: internal rotation | enrolment
  unit of measure: height of the position of the hand in the back according to anatomical landmarks; 1- lateral thigh, 2- buttock, 3- lumbosacral junction, 4- waist (L3 vertebra), 5- T12 vertebra, 6- interscapular (T7 vertebra) (worst: 1; best: 6)
Shoulder Range Of Motion: internal rotation | 3 months
  unit of measure: height of the position of the hand in the back according to anatomical landmarks; 1- lateral thigh, 2- buttock, 3- lumbosacral junction, 4- waist (L3 vertebra), 5- T12 vertebra, 6- interscapular (T7 vertebra) (worst: 1; best: 6)
Shoulder Range Of Motion: internal rotation | 6 months
  unit of measure: height of the position of the hand in the back according to anatomical landmarks; 1- lateral thigh, 2- buttock, 3- lumbosacral junction, 4- waist (L3 vertebra), 5- T12 vertebra, 6- interscapular (T7 vertebra) (worst: 1; best: 6)
Shoulder Range Of Motion: internal rotation | 12 months
  unit of measure: height of the position of the hand in the back according to anatomical landmarks; 1- lateral thigh, 2- buttock, 3- lumbosacral junction, 4- waist (L3 vertebra), 5- T12 vertebra, 6- interscapular (T7 vertebra) (worst: 1; best: 6)
Rotator cuff strength: anterior cuff | enrolment
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: anterior cuff | 3 months
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: anterior cuff | 6 months
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: anterior cuff | 12 months
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: superior cuff | enrolment
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: superior cuff | 3 months
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: superior cuff | 6 months
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: superior cuff | 12 months
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: posterior cuff | enrolment
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: posterior cuff | 3 months
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: posterior cuff | 6 months
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Rotator cuff strength: posterior cuff | 12 months
  scale 0-5 (0/5: no contraction ; 1/5: muscle contraction visible, no motion; 2/5: motion with gravity eliminated; 3/5: motion against gravity; 4/5: motion against moderate resistance; 5/5: normal muscle strength)
Apprehension test | enrolment
  examiner flexes the patient's elbow to 90° and abducts shoulder to 90°, then slowly externally rotates the patient's shoulder; the patient demonstrates apprehension during shoulder external rotation at different positions as follow: 1- early, 2- cocked position, 3- forced external rotation, 4- forced external rotation with posterior-anterior pressure (worst: 1; best: 4)
Apprehension test | 3 months
  examiner flexes the patient's elbow to 90° and abducts shoulder to 90°, then slowly externally rotates the patient's shoulder; the patient demonstrates apprehension during shoulder external rotation at different positions as follow: 1- early, 2- cocked position, 3- forced external rotation, 4- forced external rotation with posterior-anterior pressure (worst: 1; best: 4)
Apprehension test | 6 months
  examiner flexes the patient's elbow to 90° and abducts shoulder to 90°, then slowly externally rotates the patient's shoulder; the patient demonstrates apprehension during shoulder external rotation at different positions as follow: 1- early, 2- cocked position, 3- forced external rotation, 4- forced external rotation with posterior-anterior pressure (worst: 1; best: 4)
Apprehension test | 12 months
  examiner flexes the patient's elbow to 90° and abducts shoulder to 90°, then slowly externally rotates the patient's shoulder; the patient demonstrates apprehension during shoulder external rotation at different positions as follow: 1- early, 2- cocked position, 3- forced external rotation, 4- forced external rotation with posterior-anterior pressure (worst: 1; best: 4)
Subjective apprehension | enrolment
  scale 0-10 (0: no apprehension at all (= best outcome); 10: maximal apprehension (= worst outcome))
Subjective apprehension | 3 months
  scale 0-10 (0: no apprehension at all (= best outcome); 10: maximal apprehension (= worst outcome))
Subjective apprehension | 6 months
  scale 0-10 (0: no apprehension at all (= best outcome); 10: maximal apprehension (= worst outcome))
Subjective apprehension | 12 months
  scale 0-10 (0: no apprehension at all (= best outcome); 10: maximal apprehension (= worst outcome))
Relocation test | enrolment
  positive/negative; patient's shoulder is brought into 90° of abduction and maximal external rotation until the patient feels apprehension; examiner gives an antero-posterior (AP) directed pressure at the humeral head; test positive if fear of luxation is reduced after the AP pressure is applied
Relocation test | 3 months
  positive/negative; patient's shoulder is brought into 90° of abduction and maximal external rotation until the patient feels apprehension; examiner gives an antero-posterior (AP) directed pressure at the humeral head; test positive if fear of luxation is reduced after the AP pressure is applied
Relocation test | 6 months
  positive/negative; patient's shoulder is brought into 90° of abduction and maximal external rotation until the patient feels apprehension; examiner gives an antero-posterior (AP) directed pressure at the humeral head; test positive if fear of luxation is reduced after the AP pressure is applied
Relocation test | 12 months
  positive/negative; patient's shoulder is brought into 90° of abduction and maximal external rotation until the patient feels apprehension; examiner gives an antero-posterior (AP) directed pressure at the humeral head; test positive if fear of luxation is reduced after the AP pressure is applied

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Centre Epaule Coude CEPCO, Geneva
  - Hôpital La Tour, Meyrin

IPD SHARING:
Plan to Share IPD: No